CLINICAL TRIAL: NCT02589925
Title: Kombinierte Tiefe Hirnstimulation Des Nucleus Subthalamicus Und Nucleus Basalis Meynert Zur Behandlung Der Parkinson-Krankheit Mit Demenz
Brief Title: Combined Subthalamic and Nucleus Basalis Meynert Deep Brain Stimulation for Parkinson's Disease With Dementia
Acronym: Dempark-DBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DEMPARK-DBS V2.01
Record Dates: First submitted 2015-09-28; First posted 2015-10-28 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Parkinson Disease; Dementia
Keywords: deep brain stimulation; subthalamic nucleus; Nucleus basalis Meynert
MeSH Terms: conditions — Parkinson Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sham stimulation (Sham Comparator): ineffective neurostimulation of the Nucleus basalis Meynert combined with subthalamic nucleus (STN) stimulation using Vercise deep brain stimulation
  Interventions: Device: Vercise deep brain stimulation; Procedure: subthalamic nucleus (STN) stimulation; Procedure: sham stimulation
- NBM stimulation (Active Comparator): effective neurostimulation of the Nucleus basalis Meynert combined with subthalamic nucleus (STN) stimulation using Vercise deep brain stimulation
  Interventions: Device: Vercise deep brain stimulation; Procedure: subthalamic nucleus (STN) stimulation; Procedure: NBM stimulation

INTERVENTIONS:
Device: Vercise deep brain stimulation — implantation of a Vercise neurostimulation system
Procedure: subthalamic nucleus (STN) stimulation — bilateral high-frequency neurostimulation of the subthalamic nucleus using a Vercise neurostimulation system
Procedure: NBM stimulation — bilateral low-frequency neurostimulation of the subthalamic nucleus using a Vercise neurostimulation system
  Arms: NBM stimulation
Procedure: sham stimulation — ineffective neurostimulation by setting 0mA output at the Vercise neurostimulation system
  Arms: sham stimulation

SUMMARY:
Phase 1 study evaluating the safety of combined bilateral subthalamic nucleus (STN) and basal nucleus of Meynert (NBM) stimulation in treating levodopa responsive motor symptoms of Parkinsonism and cognitive dysfunction in patients with advanced Parkinson's disease having mild to moderate dementia.

DETAILED DESCRIPTION:
Combined subthalamic and Nucleus basalis Meynert Deep Brain Stimulation for Parkinson's disease with dementia DEMPARK-DBS STUDY

Indication: Parkinson's disease with mild to moderate dementia

Primary Objective: To provide a proof of safety of combined bilateral subthalamic nucleus (STN) and basal nucleus of Meynert (NBM) stimulation in treating levodopa responsive motor symptoms of Parkinsonism and cognitive dysfunction in patients with advanced Parkinson's disease having mild to moderate dementia.

Exploratory Objectives: To determine if additional NBM stimulation improves or slows progression of cognitive decline in patients with advanced Parkinson's disease having mild to moderate dementia

Test Device: Boston Scientific Corporation (BSC) Neuromodulation Vercise™ System. A neurostimulation device consisting of an implantable pulse generator (IPG), integrated rechargeable battery, two DBS leads, a splitter allowing to control four electrodes, surgical tools, and external devices (programming system, remote control, and charging system).

Device Description: The Vercise™ system IPG is a multiple independent current controlled pulse generator. The system is identical in form factor and dimensions to the commercially available 22-cc Precision Spinal Cord Stimulation II IPG. To allow the delivery of stimulation pulses to four DBS electrodes with different stimulation frequencies (100-200 Hz at the STN and 20-80 Hz at the NBM) the splitter of the Precision Spinal Cord Stimulation system will be used.

Study Design: Prospective single center Phase 1b study with double-blind randomized delayed activation of basal nucleus of Meynert neurostimulation (staggered onset design)

Planned Number of Subjects: 12 patients

Planned Number of Sites / Countries: Single center in Germany

Primary Endpoint: Safety of combined bilateral subthalamic nucleus (STN) and basal nucleus of Meynert (NBM) stimulation as determined by spontaneously reported adverse events.

Exploratory Endpoints:

* Change in global cognitive function as measured by ADAS-cog
* Change in global clinical impression as measured by ADAS-CGIC
* Change in activities of daily life as measured by ADCS-ADL and UPDRS II
* Change in neuropsychiatric symptoms as measured by BDI and Neuropsychiatric Inventory (NPI)
* Change in frontal executive function as measured by the following tests: D-KEFS verbal fluency battery, Wisconsin Card Sorting Test (modified version), Trail Making Task Part A + B, Stroop Test (Victoria Version), Symbol Digit Modalities Test
* Change in performance on the Brief Test of Attention (BTA)
* Change in apathy as measured by Starkstein Apathy Scale
* Change in motor function as assessed by UPDRS III
* Change in quality of life as assessed by PDQ39 and EQ-5d
* Change in caregiver burden/quality of life as measured by SF-36

Health Economics Endpoints:

* Gain in quality adjusted life-years (QUALY)

Method of Assigning Patients to Treatment: Eligible patients who consent to participation and have met all of the inclusion and none of the exclusion criteria will receive all of the following settings in a pre-specified randomized order for NBM neurostimulation at visit 2 :

* sham stimulation settings at 0 V, 60 µs, 20 Hz
* test stimulation at settings of 60µs, 20 Hz and individually adjusted amplitude (could be additionally verified by GUIDE visualization tool) below the threshold of adverse effects

Study Assessments:

The following assessments will be conducted to derive the study endpoints:

* ADAS-Cog
* ADAS-CGIC
* ADCS-ADL and UPDRS II
* BDI
* NPI
* Verbal Fluency from D-KEFS battery, Wisconsin Card Sorting Test (modified version), Trail Making Task Part A + B, Stroop Test (Victoria Version), Symbol Digit Modalities Test
* Brief Test of Attention
* Starkstein Apathy Scale
* UPDRS III
* Dyskinesia: Clinical Dyskinesia Rating Scale (CDRS)
* PDQ39 and EQ-5d
* Caregiver burden assessment/SF36
* Direct and indirect costs (treatment, loss of caregiver productivity, loss of patient productivity, etc.)

Study Schedule:

* Screening (0 to 4 weeks prior to inclusion)
* Presurgical baseline evaluation (motor on and off state, cognitive testing in best motor on state) (0 to 4 weeks prior to surgery)
* DBS Implant Procedure
* Postsurgical baseline evaluation (motor on and off state, cognitive testing in best motor on state) at 4±1 weeks after surgery and activation of subthalamic neurostimulation using individualized stimulation parameters after a standard monopolar review
* Visit 1 (12 weeks after activation of STN neurostimulation): motor off/on-medication + STN stimulation state, cognitive testing in motor off + STN stimulation state
* Randomization and blinded activation of NBM neurostimulation according to a 1:1 scheme
* Visit 2 (24 weeks after randomization): motor off-medication ± stimulation state, cognitive testing in motor off + STN stimulation state ± NBM stimulation state
* Activation of NBM neurostimulation in all patients
* Visit 3 (48 weeks after activation of NBM stimulation - e.g. 24 weeks after Visit 2 in the NBM neurostimulation group vs. 48 weeks): motor off -medication ± stimulation state, cognitive testing in motor off + STN stimulation state + NBM stimulation state
* Annual follow-up visit for up to 5 years after activation of NBM stimulation Required Medication Therapy Patients must be on stable doses of antiparkinsonian and antidementia medications for at least 4 weeks prior to screening assessment. Medications and dosages may be adjusted as necessary after DBS implant surgery.

Study Duration Duration of the entire trial: 2 years Duration of recruitment: 12 month Follow-Up: 9 month Statistical Analysis: 3 month Study start: 11/2015 Anticipated study end (final report): 12/2017 Duration of Treatment: 48 weeks

Statistical Methods Primary Statistical Hypothesis Sample size considerations: Emre et al NEJM 2004 found a 2.1±8.2 point improvement on the ADAS-cog with rivastigmine treatment compared to a worsening of 0.7±7.5 points with placebo after 24 weeks (baseline 23.8±10.2 points). There is currently no data to estimate treatment effect size and variability of NBM DBS. Clearly such small mean differences in combination with comparatively large standard deviations shown by the rivastigmine study are detectable with appropriate power only with sample sizes (2*125 = 250) far away from sample sizes planned for this study. But we hope to get hints to considerably larger effects for NBM DBS. Within a purely explorative analysis we will test the null hypothesis of equal mean ADAS-cog change scores from visit 1 to visit 2 for both study treatments (STN-DBS + NBM-DBS versus STN-DBS + sham-DBS) by an analysis of covariance (ANCOVA) with baseline ADAS-cog as covariate. Assuming a small to moderate correlation between baseline ADAS-cog and ADAS-cog change score from visit 1 to visit 2 a sample size of 2*5 = 10 patients ensures a power of 84% to detect a standardized mean difference of 2.0 as significant deviation from the null hypothesis of equal mean change scores for both treatments at significance level 0.05. That means we are able to detect only very large effects as significant, but this is not the main objective of this pilot study.

This study is exploratory to provide the necessary data for sample size considerations of a possible subsequent pivotal trial.

Statistical Test Method nA one-sided significance level. Sample Size Parameters nA

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of enrollment: 35 - 75 years.
2. Diagnosis of idiopathic PD with probable Parkinson's disease dementia (PDD) as defined by the MDS consensus guidelines (Emre et al., 2007)
3. Mild to moderately severe dementia as defined by a Mini-Mental State Examination (MMSE) score of 10 to 24
4. Duration of bilateral idiopathic PD: ≥5 years of motor symptoms.
5. Severity of bilateral idiopathic PD in the meds off state: modified Hoehn and Yahr stage ≥2.
6. UPDRS subset III score of ≥30 in the meds off, stim off state.
7. Levodopa must improve PD symptoms by ≥30% in a levodopa challenge test, as measured by UPDRS subset III score.
8. PDD with a symptom onset at least 2 years after first symptoms of PD
9. Be willing and able to comply with all visits and study related procedures (e.g., using the remote control, charging systems and completing the motor diary) if mentally competent or, if incompetent, their legally authorized representatives.
10. Able to understand the study requirements and the treatment procedures and to provide written informed consent before any study-specific tests or procedures are performed. If mentally incompetent, the legally authorized representative provides written informed consent

Exclusion Criteria:

1. Any significant psychiatric problems, including acute confusional state (delirium), ongoing psychosis, or clinically significant depression.
2. Any current drug or alcohol abuse.
3. Any history of recurrent or unprovoked seizures.
4. Any prior movement disorder treatments that involved intracranial surgery or device implantation.
5. A history of neurostimulation intolerance in any area of the body.
6. Any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints, including any terminal illness with survival <12 months.
7. Participation in another drug, device, or biologics trial concurrently or within the preceding 30 days. Any other trial participation should be approved by the Principal Investigators.
8. Pregnancy, breast-feeding, or lack of reliable contraception

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
safety as determined by spontaneously reported adverse events | 48 weeks
  Safety of combined bilateral subthalamic nucleus (STN) and basal nucleus of Meynert (NBM) stimulation as determined by spontaneously reported adverse events

OTHER OUTCOMES:
Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) | 48 weeks
Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADAS-CGIC) | 48 weeks
Alzheimer's Disease Co-operative Study - Activities of Daily Living Inventory (ADCS-ADL) | 48 weeks
Unified Parkinson's Disease Rating Scale section II (UPDRS II) | 48 weeks
  Unified Parkinson's Disease Rating Scale section II
Beck Depression Inventory (BDI) | 48 weeks
Neuropsychiatric Inventory (NPI) | 48 weeks
Verbal Fluency | 48 weeks
  Combined verbal fluency score from D-KEFS battery, Wisconsin Card Sorting Test (modified version), Trail Making Task Part A + B, Stroop Test (Victoria Version), Symbol Digit Modalities Test
Brief Test of Attention | 48 weeks
  auditory perception task that measures divided attention in the verbal-linguistic system
Starkstein Apathy Scale | 48 weeks
Unified Parkinson's Disease Rating Scale section III (UPDRS III) | 48 weeks
Clinical Dyskinesia Rating Scale (CDRS) | 48 weeks
EQ-5d | 48 weeks
  EQ-5D questionnaire of the EuroQol-group
Parkinson's Disease Questionnaire for quality of life (PDQ39) | 48 weeks
Caregiver burden assessment/SF36 | 48 weeks
Direct and indirect costs | 48 weeks
  cost of treatment, loss of caregiver productivity, loss of patient productivity, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Volkmann, MD, PhD, Principal Investigator — Wuerzburg University Hospital
Locations (1):
- University Hospital Würzburg, Department of Neurology, Würzburg, Germany

REFERENCES:
- [Derived] Daniels C, Steigerwald F, Capetian P, Matthies C, Malzahn U, Heuschmann PU, Volkmann J. Combined subthalamic and nucleus basalis of Meynert deep brain stimulation for Parkinson's disease with dementia (DEMPARK-DBS): protocol of a randomized, sham-controlled trial. Neurol Res Pract. 2020 Oct 19;2:41. doi: 10.1186/s42466-020-00086-w. eCollection 2020. PMID 33324941